CLINICAL TRIAL: NCT06653218
Title: Efficacy and Safety of Stellate Ganglion Block With Lidocaine Combined Platelet-rich Plasma to Treat Chronic Migraine: a Protocol of a Multi-center, Prospective, Propensity Score-matched, Cohort Analysis
Brief Title: Efficacy and Safety of Stellate Ganglion Block With Lidocaine Combined Platelet-rich Plasma to Treat Chronic Migraine
Status: Completed | Type: Observational
Sponsor: Beijing Tiantan Hospital (Other)
Collaborators: Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other); Qinghai People's Hospital (Other)
Responsible Party: Principal Investigator, Fang Luo, Director of Department of pain management, Beijing Tiantan Hospital
Other Study IDs: KY-2023-263-03-06
Record Dates: First submitted 2024-10-20; First posted 2024-10-22 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Platelet-rich Plasma; Chronic Migraine
Keywords: Platelet-rich Plasma; Chronic Migraine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- PRP+Lidocaine group: Patients will be placed in the supine position, with slightly excessive neck extension to receive stellate ganglion block (SGB). And 2.5 ml of PRP combined with 2.5 ml of 1.0% lidocaine will be injected slowly into the ipsilateral stellate ganglion under the guide of ultrasound visualization technology
  Interventions: Other: No interventions
- Lidocaine group: Patients will be placed in the supine position, with slightly excessive neck extension to receive stellate ganglion block (SGB). And 5 ml of 1.0% lidocaine will be injected slowly into the ipsilateral stellate ganglion under the guide of ultrasound visualization technology
  Interventions: Other: Not have interventions

INTERVENTIONS:
Other: No interventions — It is a observational study
  Groups: PRP+Lidocaine group
Other: Not have interventions — It is a observational study
  Groups: Lidocaine group

SUMMARY:
This is a multicenter, prospective, observational, propensity score matching, cohort, and assessor-blinded study designed to compare the effectiveness and safety of lidocaine combined Platelet-rich plasma (PRP) acting on SGB versus lidocaine alone acting on SGB in patients with CM.

DETAILED DESCRIPTION:
Chronic migraine (CM) is a disabling disease that causes serious physical and emotional consequences. Previous studies had suggested the efficacy of stellate ganglion block (SGB) with lidocaine in the treatment of CM. However, the side effects related to repeated procedures limit its applications. Platelet-rich plasma (PRP) as an intervention treatment for chronic pain, has shown promising results to alleviate headache within the distribution range of the greater occipital nerve after trauma. So far, there has not been any report on PRP combined with lidocaine acting on SGB for CM. the investigators will conduct this multicenter, prospective, observational, propensity score matching, cohort, and assessor-blinded study to evaluate the efficacy and safety of lidocaine combined PRP acting on SGB versus lidocaine alone acting on SGB in patients with CM

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18 to 75 years;
2. BMI between 15 and 35 kg/m2 ;
3. Diagnosed with CM in accordance with the International Classification of Headache Disorders, 3rd Edition (ICHD-3) criteria (Headache Classification Committee of the International Headache Society (IHS) The International Classification of Headache Disorders, 3rd edition. Cephalalgia. 2018 Jan;38(1):1-211);
4. Visual Analogue Scale (VAS; range, 0-10; 0 = no pain and 10 = worst possible pain; higher scores indicate more severe pain) score≥4;
5. Scheduled for lidocaine acting on SGB treatment for CM；
6. Signed informed consent.

Exclusion Criteria:

1. Previously received SGB treatment;
2. Combined with other types of headaches;
3. Platelet count <105*109/L, use of anticoagulants or antiplatelet agent, coagulation disorders or bleeding disorders;
4. Infection or mass near the puncture site;
5. A history of other neurological disorders;
6. A history of severe cardiopulmonary, hepatic or renal dysfunction;
7. A history of psychological disorders;
8. A history of narcotic drug abuse;
9. Changes in neck anatomic structure caused by radiotherapy or surgery;
10. A history of allergies to any research drugs;
11. Pregnancy or lactation period.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: We speculate that the reduction value in monthly headache days after PRP combined lidocaine acting on SGB is expected to 2.0, and the standard deviation (SD) for the PRP group is 9.0. Assuming a 20% rate of loss to follow-up and an additional 40% loss after PSM, a total of 200 participants will provide 90% power to use a 0.05 two tailed alpha to detect the significant difference in the monthly headache days. Three participating centers will compete to enroll patients.
Sampling Method: Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2024-10-20 (Actual); Primary Completion 2025-06-30 (Actual); Study Completion 2025-09-30 (Actual)

PRIMARY OUTCOMES:
the change from baseline in mean headache days across the 1-month follow-up period. | 1-month period
  the change from baseline in mean headache days across the 1-month follow-up period.

SECONDARY OUTCOMES:
50% responder rate | at weeks 4, 8, 12.
  the proportion of patients who achieved a ≥50% reduction in monthly headache days.
Mean VAS score during headache attack | at baseline and weeks 4, 8, 12.
  evaluation of the average severity of headache days
Analgesic consumption | at baseline and weeks 4, 8, 12.
  including the number of days, the specific drug used, and the dose of drugs.
Patient satisfaction (PS) scores | at weeks 4, 8, 12.
  It ranges from 0 to 10 points, and 0 indicates unsatisfactory, while 10 points indicate very satisfactory.A higher scores mean a better satisfaction
Headache impact test version 6 (HIT-6) | at baseline and weeks 4, 8,12.
  a six-item survey that assesses the adverse impact of headaches on social, role and cognitive functioning, vitality, and psychological distress.A larger score reflects a greater adverse impact. It ranges from 36 to 78, where a higher score indicates a greater impact of headache on the daily life of the respondent
Migraine disability assessment (MIDAS) scores | at baseline and weeks 4, 8, 12.
  to evaluate headache-related disability using 4-week recall, and is associated with headache frequency and average pain score.The score ranges from 0 to 270. Higher scores indicate greater disability caused by headaches with scores of 21 or greater considered severe.
Hospital anxiety and depression scale (HADS) scores | at baseline and weeks 4, 8, 12.
  a 14-item self-report instrument used to screen for anxiety and depression separately.The range of the scale is 0 to 21, with scores of 8 to 10 being indicative of a probable risk of anxiety or depression, whereas scores of 11 to 21 indicate a high risk of anxiety or depression
Pittsburgh sleep quality index (PSQI) scores | at baseline and weeks 4, 8, 12
  a 19-item self-report instrument that comprises 7 components used to assess quality of sleep. The range of the scale is 0 to 21,with a higher score indicating more severe sleep disturbances.
Adverse events | at day 0, 1, weeks 1, 4, 8, 12
  9. including SGB-related complication and medication-related complication.

CONTACTS AND LOCATIONS:
Overall Officials: Fang Luo, M.D., Principal Investigator — Beijing Tiantan Hospital
Locations (1):
- Fang Luo, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No
not yet decided